CLINICAL TRIAL: NCT06685198
Title: The Impact of Different Titration Endpoints of Propofol on Hemodynamics and Stress During the Induction Phase of General Anesthesia
Brief Title: Observation on Administration of Propofol at Different Titration Endpoints
Acronym: OAPDTE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SanQing Jin (Other)
Responsible Party: Sponsor-Investigator, SanQing Jin, professor, Sixth Affiliated Hospital, Sun Yat-sen University
Organization: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2024ZSLYEC-457
Record Dates: First submitted 2024-11-09; First posted 2024-11-12 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Anesthesia, General; Hemodynamics
Keywords: titration of propofol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group O (Experimental): Titrated administration of propofol to an OAA/S score of 1 as the endpoint.
  Interventions: Procedure: Titrated administration of propofol to an OAA/S score of 1 as the endpoint
- Group T (Experimental): Titrated administration of propofol to an OAA/S score of 2 as the endpoint.
  Interventions: Procedure: Titrated administration of propofol to an OAA/S score of 2 as the endpoint
- Group B (Active Comparator): Titrated administration of propofol to a BIS value ≤ 60 as the endpoint.
  Interventions: Procedure: Titrated administration of propofol to a BIS value ≤ 60 as the endpoint

INTERVENTIONS:
Procedure: Titrated administration of propofol to an OAA/S score of 1 as the endpoint — Propofol is titrated at a rate of 0.5 mg/kg/min to achieve an OAA/S score of 1, followed by a maintenance dose of 2-4 mg/kg/h, concurrently with remifentanil 2 ug/kg and rocuronium 0.6 mg/kg for anesthesia induction.
  Arms: Group O
Procedure: Titrated administration of propofol to an OAA/S score of 2 as the endpoint — Propofol is titrated at a rate of 0.5 mg/kg/min to achieve an OAA/S score of 2, followed by a maintenance dose of 2-4 mg/kg/h, concurrently with remifentanil 2 ug/kg and rocuronium 0.6 mg/kg for anesthesia induction.
  Arms: Group T
Procedure: Titrated administration of propofol to a BIS value ≤ 60 as the endpoint — Propofol is titrated at a rate of 0.5 mg/kg/min to achieve a BIS value ≤ 60, followed by a maintenance dose of 2-4 mg/kg/h, concurrently with remifentanil 2 ug/kg and rocuronium 0.6 mg/kg for anesthesia induction.
  Arms: Group B

SUMMARY:
Propofol has a rapid onset and short duration of action, making it widely used for induction of general anesthesia. However, its prominent drawback is circulatory depression. Our research team previously proposed an individualized dosing method for the titration of propofol. We then compared the effects of different titration rates of propofol on hemodynamics and stress during general anesthesia induction. It was found that the incidence of hypotension during the induction period was lower in the 0.5 mg/kg/min group, with lower stress levels and faster postoperative recovery. However, this group still had a 25.3% incidence of hypotension. Therefore, we plan to further study the differences in hemodynamics, depth of anesthesia, stress response, and postoperative recovery in three groups of patients induced with a constant infusion rate of propofol at 0.5 mg/kg/min titrated to an OAA/S score of 1, an OAA/S score of 2, and BIS ≤ 60, combined with remifentanil 2 μg/kg. This study aims to explore the appropriate propofol titration endpoint during general anesthesia induction to maintain stable perioperative haemodynamics and achieve rapid postoperative recovery.

DETAILED DESCRIPTION:
Propofol can rapidly induce sleep in patients, creating favorable conditions for tracheal intubation, and is widely used for the induction of general anesthesia for tracheal intubation. However, its prominent drawback is circulatory depression. In clinical practice, propofol is still commonly administered for the induction of general anesthesia as a single intravenous bolus at the recommended dose (2-2.5 mg/kg). This method does not take into account individual differences and easily causes hypotension. In addition, target-controlled infusion under BIS monitoring is used in some cases. However, this approach requires high standards of equipment, has limited clinical applicability, and there is still controversy over whether the targetcontrolled model accurately reflects the concentration of propofol in blood or brain tissue.A 2020 retrospective study by Eric Y. et al. showed that the anesthetic induction dose of propofol for elderly patients was not adequately adjusted according to recommendations, resulting in an excessive actual dose. There are also studies on titrated administration of propofol, but the endpoints for titrated administration are still unclear.

Hypotension during the induction period has been identified as an independent predictor of adverse clinical outcomes. Early studies suggested that a mean arterial pressure (MAP) of <50-55 mmHg or a reduction in systolic blood pressure (SBP) or MAP by more than 40-50% from baseline can cause organ dysfunction.As research into the dangers of hypotension deepens, the minimum value that hypotension may cause damage is continuously increasing, and the harm brought by mild hypotension is increasingly being taken seriously. The impact of induced hypotension during the induction period on patients is related to the severity, duration of hypotension, and the patient's baseline condition.

Hypotension during the induction period of anesthesia is largely preventable and should be prevented. Therefore, finding appropriate endpoints for propofol titration can reduce the incidence of hypotension during the induction period, which is of ignificant significance for improving the prognosis of surgical patients.

Common methods for monitoring the depth of anesthesia during the induction period of general anesthesia include observer-based evaluations, such as the Observer's Assessment of Alertness/Sedation (OAA/S) score, and machinebased evaluations, such as the Bispectral Index (BIS) score.

The OAA/S score is a commonly used clinical observation tool that is simple and convenient to operate, requiring no additional equipment. It mainly assesses the depth of sedation by giving verbal commands and tactile stimuli to the patient. Various studies have shown that it correlates closely with machinebased indices for monitoring the depth of anesthesia, such as the BIS and the Index of Consciousness (IOC). As a straightforward, cost-effective method for monitoring the depth of anesthesia, the OAA/S score is closely related to clinical manifestations and is particularly suitable for monitoring the depth of anesthesia during the induction period.

BIS (Bispectral Index) is a quantitative electroencephalogram (EEG) parameter that transforms the frequency, amplitude, and phase characteristics of the EEG through fast Fourier transformation, providing a numerical value between 0 (suppressed state) and 100 (awake state) to quantify different depths of anesthesia. However,the BIS value is influenced by various factors;neuromuscular blockers can interfere with BIS readings,while esmolol and epinephrine can increase BIS readings. Some studies have shown that BIS monitoring does not reduce intraoperative awareness and the amount of anesthetic agents used.Since the calculation and analysis of EEG data require time, there is a delay of approximately 30.09 ± 18.73 seconds in monitoring the depth of anesthesia with BIS. Therefore, BIS has limitations in monitoring the depth of anesthesia.

Currently, many studies use BIS for monitoring the depth of anesthesia during surgery. Some research has shown that titrated administration of propofol based on BIS monitoring (40-60) during the induction period of general anesthesia does not differ in propofol dosage and incidence of hypotension compared to conventional single-dose administration. This prompts the critical inquiry: Is BIS an appropriate measure for assessing the depth of anesthesia during the induction period of general anesthesia? In the first phase of our previous research, we proposed an individualized dosing strategy for slow constant-rate infusion of propofol, using an OAA/ S score of 1 as the titration endpoint. Through a randomized controlled trial comparing the hemodynamic effects of slow infusion of propofol (1 mg/kg/ min) versus the traditional single-dose administration (2 mg/kg, 250 mg/min) during the induction period of general anesthesia, we found that the titrated administration of propofol not only mitigated the extent of blood pressure reduction, but also decreased the overall amount of propofol required during the induction phase.

In the second phase, we further designed a randomized controlled doubleblind trial to explore appropriate titration infusion rate. We studied the effects of titrated induction at infusion rates of 2 mg/kg/min, 1 mg/kg/min, and 0.5 mg/ kg/min on hemodynamics, brain activity, blood concentration of propofol, and stress response. We found that all three titration methods achieved the required depth of anesthesia for tracheal intubation. The 0.5 mg/kg/min group had a more stable blood concentration curve of propofol, lower incidence of hypotension and low BIS during the induction period, lower stress levels, and shorter recovery time after surgery.Based on the research, we found that the 0.5 mg/kg/min group still had a 25.3% incidence of hypotension, with the proportion of cases with mean arterial pressure <65 mmHg as high as 47.3%. Therefore, we hypothesize that adopting an OAA/S score of 2 as the titration endpoint might be more reasonable.

This study aims to compare the differences between using different OAA/S scores and BIS value for guiding titrated administration of propofol during the induction period of general anesthesia. We seek to explore a reasonable and feasible titration endpoint for propofol to reduce the incidence of hypotension during induction, maintain stable perioperative vital signs, and facilitate rapid postoperative recovery.

The protocol involves a planned enrollment of 258 patients scheduled for surgery under tracheal intubation and general anesthesia. They will be randomly divided into 3 groups of 86 patients each according to a random number table. During the induction of anesthesia, the pump operator will adjust propofol at a rate of 0.5 mg/kg/min based on the envelope group (Groups O, T, B), titrating to the respective endpoints (OAA/S score of 1, OAA/S score of 2, BIS ≤ 60). Propofol will then be adjusted to a maintenance dose of 2-4 mg/ kg/h, combined with remifentanil 2 ug/kg and rocuronium 0.6 mg/kg. Tracheal intubation will commence 2 minutes after muscle relaxant administration. Researchers will observe hemodynamic changes and EEG activity throughout the process, adjusting medications to maintain stable hemodynamics as much as possible.

After confirming the successful tracheal intubation, the investigators will give participants machine-controlled ventilation, and the total intravenous anesthesia(TIVA) will be given with propofol, remifentanil, and cis-atracurium. During the operation, remifentanil will be injected with a constant rate of 0.2ug/ kg/min, and propofol will be injected with a fluctuating rate of 2-8mg/kg/h (the pump injection rate will be adjusted according to blood pressure and BIS, and the rate of remifentanil can be adjusted if necessary) to maintain BIS between 40-60.Fluid therapy will be performed according to the participants' hemodynamics and intraoperative conditions. After extubation, participants will be sent to the postoperative recovery room; a follow-up visit will be performed the next day,and a telephone return visit will be performed on the 30th day.

Researchers recorded the preoperative day Recovery Quality (Qor-15) scores for each participant, preoperative anxiety (VAS) scores upon entry; maximum and minimum blood pressure during anesthesia induction, BIS values corresponding to different OAAS scores and the lowest BIS value during induction. and corresponding times of propofol titration to OAA/S scores; total doses of propofol, remifentanil, rocuronium, and vasopressors during induction; pupil size and reflex assessments at four time points (before sleep, at titration endpoint, before intubation, after intubation); auditory evoked potentials (AEP) and electroencephalogram monitoring before propofol administration and at titration endpoint; blood draws at three time points (pre-induction, titration endpoint, 30 seconds post-tracheal intubation) for glucose and stress indicators catecholamines (epinephrine, norepinephrine); postoperative assessment of intraoperative awareness and postoperative memory, and cardiovascular events within 30 days postoperatively recorded with Recovery Quality (Qor-15) scores.

Parameters recorded during induction include systolic blood pressure (SBP), diastolic blood pressure (DBP), mean arterial pressure (MAP), heart rate (HR), BIS value, cardiac function parameters [heart rate variability (HRV), stroke volume (SV), stroke index (SVI), cardiac output (CO), cardiac index (CI)), oxygen delivery parameters (oxygen delivery (DO2), oxygen delivery index (DO2I)], peripheral vascular resistance parameters [systemic vascular resistance (SVR), systemic vascular resistance index (SVRI)], volume parameters [stroke volume variation (SVV), pulse pressure variation (PPV), increase in stroke volume (SV)], auditory evoked potential parameters [brain stem auditory evoked potentials (BAEP):latency and amplitude of waves III, V; middle latency auditory evoked potentials (MLAEP): latency and amplitude of waves Pa, Nb], and EEG parameters (power spectrum of β, α, θ, and σ brain waves).

Blinded design: After assigning intervention measures, blinding is implemented for subjects and researchers (principal investigator, main anesthesiologist, postanesthesia care unit physician, postoperative follow-up physician).The principal investigator of the research team generates allocation numbers and recruits participants. During induction, the specific grouping of anesthesia patients is unknown, and each patient receives a complete assessment of OAA/S scores.

The research team instructs the anesthesiologist in charge of adjusting the infusion pump to: collect experimental envelopes from the research assistant in advance, set up the infusion pump, position the pump away from the primary observers and main anesthesiologist, and adjust propofol administration based on grouping, combined with assessments by the principal investigator or BIS values. Propofol administration is stopped upon reaching the titration endpoint, followed by maintenance doses, and administration of remifentanil and rocuronium is given. The doses of propofol and induction times are recorded. During induction, the anesthesiologist follows instructions from the principal investigator to administer additional vasopressors or propofol and does not participate in postoperative follow-up tasks.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-60 years.
2. Elective surgery with planned endotracheal intubation under general anesthesia.
3. ASA classification of I or II,with heart function classified as 1 or 2.
4. Body Mass Index (BMI) 18-30 kg/m².

Exclusion Criteria:

1. Severe cardiac, pulmonary, hepatic, or renal diseases (heart function classification greater than 3 / respiratory failure / liver failure / renal failure).
2. Malignant arrhythmias: atrial flutter, atrial fibrillation, atrioventricular block, frequent ventricular premature beats, multifocal ventricular premature beats, ventricular premature beats R on T, ventricular flutter, and ventricular fibrillation.
3. Expected difficulty with intubation, hypoalbuminemia, hypertension, or diabetes mellitus.
4. Patients with a high risk of aspiration due to a full stomach, gastrointestinal obstruction, or pregnancy.
5. Patients with schizophrenia, epilepsy, Parkinson's disease, intellectual disabilities, etc.
6. Alcohol abusers or those who have been using sedatives or analgesics long-term.
7. Allergic to propofol or its emulsion.
8. Currently participating in a clinical trial that conflicts with this study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 258 (Estimated)
Dates: Start 2025-02-20 (Estimated); Primary Completion 2025-06-20 (Estimated); Study Completion 2025-08-20 (Estimated)

PRIMARY OUTCOMES:
Incidence of a 30% decrease in MAP | During the procedure of anesthesia induction
  Incidence of a 30% decrease in MAP during induction with three different titration endpoints

SECONDARY OUTCOMES:
Proportion of cases with MAP < 65 mmHg | During the procedure of anesthesia induction
  Proportion of cases with MAP < 65 mmHg during induction in three groups
Anesthesia depth | During the procedure of anesthesia induction
  Anesthesia depth during induction in three groups (BIS values,pupil size and reaction to light,EEG patterns,auditory evoked potentials)
Tracheal intubation conditions | After finish intubation
  Differences of the tracheal intubation conditions of patients among the three groups
Blood glucose | During the procedure of anesthesia induction
  Blood glucose before induction,at the end of titration,and 30 seconds after endotracheal intubation in three groups
Stress hormones | During the procedure of anesthesia induction
  Stress indicators (catecholamines: adrenaline,noradrenaline) before induction,at the end of titration,and 30 seconds after endotracheal intubation in three groups.
Mean Arterial Pressure（MAP） | During the procedure of anesthesia induction
  Changes in MAP during induction in three groups
Heart Rate(HR) | During the procedure of anesthesia induction
  Changes in HR during induction in three groups
Cardiac Index(CI) | During the procedure of anesthesia induction
  Changes in CI during induction in three groups
Stroke Volume Index(SVI) | During the procedure of anesthesia induction
  Changes in SVI during induction in three groups
Systemic Vascular Resistance Index(SVRI) | During the procedure of anesthesia induction
  Changes in SVRI during induction in three groups
Propofol dosage | During the procedure of anesthesia induction
  Propofol dosage during induction in three groupsThe dosage of propofol (Reach the end of the titration, complete the tracheal intubation, and complete the operation) and usage of vasoactive drugs in the three groups
Induction time | After finish operation
  Induction time in the three groups
Recovery time | From surgery completion to first recovery
  Postoperative recovery time
Length of hospital stay after surgery | From surgery completion to actual hospital discharge,assessed up to 30 days
  Hospital stay time from operation completion to actual hospital discharge
Cognitive and memory function | Postoperative Day 1 and Day 30
  Modified Brice Questionnaire,Three-Word Recall Test,AD-8 Self-Assessment for Cognitive Impairment
Recovery quality | Preoperative Day 1 and postoperative Day 1 and Day 30
  Postoperative recovery score using 15-item quality of recovery scoring system(QoR-15)
The occurrence of important cardiovascular events | Within 30 days after surgery
  The occurrence of important cardiovascular events during the perioperative period

CONTACTS AND LOCATIONS:
Overall Officials: SanQing Jin, MD, Principal Investigator — The Sixth Affiliated Hospital, Sun Yat-sen University
Locations (1):
- the Sixth Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rusch D, Arndt C, Eberhart L, Tappert S, Nageldick D, Wulf H. Bispectral index to guide induction of anesthesia: a randomized controlled study. BMC Anesthesiol. 2018 Jun 15;18(1):66. doi: 10.1186/s12871-018-0522-8. PMID 29902969
- [Background] Hino H, Matsuura T, Kihara Y, Tsujikawa S, Mori T, Nishikawa K. Comparison between hemodynamic effects of propofol and thiopental during general anesthesia induction with remifentanil infusion: a double-blind, age-stratified, randomized study. J Anesth. 2019 Aug;33(4):509-515. doi: 10.1007/s00540-019-02657-x. Epub 2019 Jun 21. PMID 31228006
- [Background] Chen EY, Michel G, Zhou B, Dai F, Akhtar S, Schonberger RB. An Analysis of Anesthesia Induction Dosing in Female Older Adults. Drugs Aging. 2020 Jun;37(6):435-446. doi: 10.1007/s40266-020-00760-3. PMID 32300966
- [Background] Green RS, Butler MB. Postintubation Hypotension in General Anesthesia: A Retrospective Analysis. J Intensive Care Med. 2016 Dec;31(10):667-675. doi: 10.1177/0885066615597198. Epub 2016 Jul 7. PMID 26721639
- [Background] Jor O, Maca J, Koutna J, Gemrotova M, Vymazal T, Litschmannova M, Sevcik P, Reimer P, Mikulova V, Trlicova M, Cerny V. Hypotension after induction of general anesthesia: occurrence, risk factors, and therapy. A prospective multicentre observational study. J Anesth. 2018 Oct;32(5):673-680. doi: 10.1007/s00540-018-2532-6. Epub 2018 Jul 19. PMID 30027443
- [Background] Hallqvist L, Martensson J, Granath F, Sahlen A, Bell M. Intraoperative hypotension is associated with myocardial damage in noncardiac surgery: An observational study. Eur J Anaesthesiol. 2016 Jun;33(6):450-6. doi: 10.1097/EJA.0000000000000429. PMID 26950081
- [Background] Walsh M, Devereaux PJ, Garg AX, Kurz A, Turan A, Rodseth RN, Cywinski J, Thabane L, Sessler DI. Relationship between intraoperative mean arterial pressure and clinical outcomes after noncardiac surgery: toward an empirical definition of hypotension. Anesthesiology. 2013 Sep;119(3):507-15. doi: 10.1097/ALN.0b013e3182a10e26. PMID 23835589
- [Background] Sun LY, Chung AM, Farkouh ME, van Diepen S, Weinberger J, Bourke M, Ruel M. Defining an Intraoperative Hypotension Threshold in Association with Stroke in Cardiac Surgery. Anesthesiology. 2018 Sep;129(3):440-447. doi: 10.1097/ALN.0000000000002298. PMID 29889106
- [Background] Gregory A, Stapelfeldt WH, Khanna AK, Smischney NJ, Boero IJ, Chen Q, Stevens M, Shaw AD. Intraoperative Hypotension Is Associated With Adverse Clinical Outcomes After Noncardiac Surgery. Anesth Analg. 2021 Jun 1;132(6):1654-1665. doi: 10.1213/ANE.0000000000005250. PMID 33177322
- [Background] Ahuja S, Mascha EJ, Yang D, Maheshwari K, Cohen B, Khanna AK, Ruetzler K, Turan A, Sessler DI. Associations of Intraoperative Radial Arterial Systolic, Diastolic, Mean, and Pulse Pressures with Myocardial and Acute Kidney Injury after Noncardiac Surgery: A Retrospective Cohort Analysis. Anesthesiology. 2020 Feb;132(2):291-306. doi: 10.1097/ALN.0000000000003048. PMID 31939844
- [Background] Chernik DA, Gillings D, Laine H, Hendler J, Silver JM, Davidson AB, Schwam EM, Siegel JL. Validity and reliability of the Observer's Assessment of Alertness/Sedation Scale: study with intravenous midazolam. J Clin Psychopharmacol. 1990 Aug;10(4):244-51. PMID 2286697
- [Background] Kasuya Y, Govinda R, Rauch S, Mascha EJ, Sessler DI, Turan A. The correlation between bispectral index and observational sedation scale in volunteers sedated with dexmedetomidine and propofol. Anesth Analg. 2009 Dec;109(6):1811-5. doi: 10.1213/ANE.0b013e3181c04e58. PMID 19923507
- [Background] Schick A, Driver B, Moore JC, Fagerstrom E, Miner JR. Randomized Clinical Trial Comparing Procedural Amnesia and Respiratory Depression Between Moderate and Deep Sedation With Propofol in the Emergency Department. Acad Emerg Med. 2019 Apr;26(4):364-374. doi: 10.1111/acem.13548. Epub 2018 Sep 24. PMID 30098230
- [Background] Schuller PJ, Newell S, Strickland PA, Barry JJ. Response of bispectral index to neuromuscular block in awake volunteers. Br J Anaesth. 2015 Jul;115 Suppl 1:i95-i103. doi: 10.1093/bja/aev072. PMID 26174308
- [Background] Ferreira AL, Mendes JG, Nunes CS, Amorim P. [Evaluation of Bispectral Index time delay in response to anesthesia induction: an observational study]. Braz J Anesthesiol. 2019 Jul-Aug;69(4):377-382. doi: 10.1016/j.bjan.2019.03.008. Epub 2019 Jul 29. PMID 31371175
- [Background] Choi SH, Kim CS, Kim JH, Kim BS, Kim EM, Min KT. A single dose of esmolol blunts the increase in bispectral index to tracheal intubation during sevoflurane but not desflurane anesthesia. J Neurosurg Anesthesiol. 2009 Jul;21(3):214-7. doi: 10.1097/ANA.0b013e3181a41e69. PMID 19542998
- [Background] Avidan MS, Zhang L, Burnside BA, Finkel KJ, Searleman AC, Selvidge JA, Saager L, Turner MS, Rao S, Bottros M, Hantler C, Jacobsohn E, Evers AS. Anesthesia awareness and the bispectral index. N Engl J Med. 2008 Mar 13;358(11):1097-108. doi: 10.1056/NEJMoa0707361. PMID 18337600
- [Background] Chen L, Lu K, Luo T, Liang H, Gui Y, Jin S. Observer's Assessment of Alertness/Sedation-based titration reduces propofol consumption and incidence of hypotension during general anesthesia induction: A randomized controlled trial. Sci Prog. 2021 Oct;104(4):368504211052354. doi: 10.1177/00368504211052354. PMID 34825617
- [Background] Bijker JB, Persoon S, Peelen LM, Moons KG, Kalkman CJ, Kappelle LJ, van Klei WA. Intraoperative hypotension and perioperative ischemic stroke after general surgery: a nested case-control study. Anesthesiology. 2012 Mar;116(3):658-64. doi: 10.1097/ALN.0b013e3182472320. PMID 22277949